CLINICAL TRIAL: NCT07291622
Title: Effect of a Synchrony-Optimized Non-Invasive Ventilation Education Program on Intensive Care Unit Patients' Outcomes: A Randomized Clinical Trial Protocol
Brief Title: Synchrony-Optimized Non-Invasive Ventilation Education Program and ICU Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sogand Sarmadi, Principal Investigator, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IR.SBMU.RETECH.REC.1404.593
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Ventilator Associated Events; Asynchrony, Patient-Ventilator; Intensive Care (ICU); Noninvasive Ventilation
Keywords: Non-Invasive Ventilation; Patient-Ventilator Synchrony; Intensive Care Unit (ICU); Anxiety and Depression; Randomized Clinical Trial; Patient Comfort
MeSH Terms: conditions — Patient-Ventilator Asynchrony; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYNC-NIV (Experimental): The intervention will consist of a structured two-session synchrony-optimized NIV education program designed to improve patient-ventilator interaction and reduce NIV-related complications. In the first 20-40-minute session, patients will be taught the ventilator's inspiratory and expiratory cycles and will practice synchronizing their breathing with the device through guided diaphragmatic exercises and real-time feedback until they demonstrate stable synchrony. The second 45-60-minute session, delivered 18-24 hours later, will provide supplementary training on proper mask selection and fixation, prevention of common NIV complications, leak reduction techniques, equipment maintenance, advanced breathing exercises, and basic ventilator monitoring and alarm management. An educational booklet summarizing all essential topics will be provided to support ongoing adherence and self-management.
  Interventions: Other: SYNC-NIV
- Control Group (No Intervention): Standard care will include regular education on the ICU environment, basic intensive care processes, the use of monitoring devices, ICU rules, effective communication with critically ill patients, and basic principles of patient care.

INTERVENTIONS:
Other: SYNC-NIV — The intervention will include two educational sessions to improve patient-ventilator synchrony and NIV management. The first session will teach patients about the ventilator's breathing cycles and train them to coordinate their breathing using visual aids and hands-on practice with real-time feedback. Competency will be assessed by their ability to maintain synchrony with minimal mask leak. The second session, held 18-24 hours later, will cover mask fitting, prevention of common complications, leak reduction, equipment care, advanced breathing exercises, and basic ventilator alarm management. Communication and relaxation techniques will also be taught, and patients will receive a booklet summarizing the key information.
  Arms: SYNC-NIV

SUMMARY:
The aim of this clinical trial is to find out whether a synchrony-optimized education program for non-invasive ventilation (NIV) can help ICU patients use their ventilator more effectively and improve their comfort, symptoms, and psychological well-being.

Researchers want to answer these main questions:

Can a structured two-session NIV education program help patients use their ventilator more regularly and for longer periods?

Does this type of training reduce anxiety, depression, and respiratory symptoms?

Can synchrony training improve patients' comfort and reduce NIV-related problems such as mask leaks or sleep disturbances?

Is this program more effective than the routine ICU education normally provided?

What Will Happen in the Study

Adults (18+) who are receiving NIV in the ICU will participate in this study.

Participants will be randomly assigned to one of two groups:

Intervention Group: Will receive the SYNC-NIV education program, consisting of:

One hands-on session (20-40 minutes) teaching patients how to synchronize their breathing with the ventilator

One supplementary session (45-60 minutes) covering mask management, preventing complications, reducing leaks, breathing exercises, equipment care, and alarm handling

An educational booklet for continued support

Control Group: Will receive the standard ICU education normally provided about the ICU environment, general care, communication, and monitoring.

All participants will be evaluated at three times:

before the intervention, the day after the program ends, and one week later.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age
* Admitted to the ICU for at least 24 hours
* Anticipated to be hospitalized for more than one week
* Receiving NIV treatment for any underlying condition
* Capable of learning
* Proficient in the Persian language

Exclusion Criteria:

* Patients with Richmond Agitation-Sedation Scale (RASS) scores of +4 or -5
* Patients with cognitive disorders
* Patients with neurological disorders
* Patients with anxiety disorders
* Patients whose condition deteriorates, making continued cooperation impossible
* Patients unable to participate in educational sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-12-19 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
NIV Usage | Baseline, the day after SYNC-NIV program completion, and 1 week after program completion
  Adherence data, including daily NIV usage, will be retrieved from the NIV machine. Adherence will be defined as more than 4 hours of nighttime use for more than 70% of days until study completion or a mean daily use of more than 5 hours.

SECONDARY OUTCOMES:
Anxiety and Depression | Baseline, the day after SYNC-NIV program completion, and 1 week after program completion
  Levels of anxiety and depression will be assessed using the Hospital Anxiety and Depression Scale (HADS), a 14-item self-report instrument divided into two subscales: anxiety (HADS-A) and depression (HADS-D), each comprising seven items. Participants will rate each item on a 4-point scale (0-3), yielding subscale scores ranging from 0 to 21. Scores for both subscales will be interpreted as follows: 0-7 indicating no symptoms, 8-10 mild, 11-14 moderate, and 15-21 severe. The internal consistency of the anxiety subscale (HADS-A) and depression subscale (HADS-D) will have been demonstrated with Cronbach's alpha coefficients of 0.820 and 0.807, respectively. The Persian version of the HADS will have shown good reliability and validity in clinical populations. Montazeri et al. (2003) will have found it acceptable by 99% of patients, with Cronbach's alpha of 0.78 for anxiety and 0.86 for depression subscales.
Respiratory Symptoms, Sleep Quality, and NIV-Associated Adverse Events | Baseline, the day after SYNC-NIV program completion, and 1 week after program completion
  Respiratory Symptoms, Sleep Quality, and NIV-Associated Adverse Events The S3-NIV Questionnaire will be a self-administered tool that includes 11 questions, all scored by patients on a 5-point Likert scale that ranges from 0 to 4 (0 = always true; 1 = mostly true; 2 = sometimes true; 3 = mostly untrue; 4 = completely untrue), based on their experiences over the previous four weeks. To calculate the overall score, the average of all completed items will be multiplied by 2.5. A score of zero will reflect the highest degree of disease impact, whereas a score of ten will reflect the lowest. Two subscale scores may also be derived: the "Respiratory Symptoms" sub score will be computed by averaging responses to items 1, 4, 5, 6, and 7 and multiplying by 2.5, while the "Sleep & Side Effects" sub score will be based on the average of items 2, 3, 8, 9, 10, and 11, also multiplied by 2.5.
Comfort | Baseline, the day after SYNC-NIV program completion, and 1 week after program completion
  To evaluate participants' comfort levels, the Visual Analog Scale (VAS) will be employed. The VAS will be a widely used, reliable, and sensitive instrument for assessing subjective experiences such as comfort (6). It typically will consist of a 10-centimeter horizontal line anchored by two extremes, for example, "no discomfort" on the left end (score 0) and "worst possible discomfort" on the right end (score 10). Participants will mark a point along the line that best represents their perceived level of comfort. The simplicity, sensitivity, and ease of administration of the VAS will make it a preferred tool in both clinical and research settings for quantifying subjective states.

IPD SHARING:
Plan to Share IPD: Undecided